CLINICAL TRIAL: NCT01734785
Title: A Phase III, Randomised, Double-blind, Parallel Group, 24 Week Study to Evaluate Efficacy and Safety of Once Daily Empagliflozin 10 mg and 25 mg Compared to Placebo, All Administered as Oral Fixed Dose Combinations With Linagliptin 5 mg, in Patients With Type 2 Diabetes Mellitus and Insufficient Glycaemic Control After 16 Weeks Treatment With Linagliptin 5 mg Once Daily on Metformin Background Therapy.
Brief Title: Safety and Efficacy of the Combination of Empagliflozin and Linagliptin Compared to Linagliptin Alone Over 24 Weeks in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1275.9; 2012-002270-31 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-11-16; First posted 2012-11-28 (Estimated); Results first posted 2016-04-18 (Estimated); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin; empagliflozin

ARMS (3):
- Linagliptin (Active Comparator): 5 mg once daily
  Interventions: Drug: Linagliptin; Drug: Empagliflozin placebo + Linagliptin placebo
- Empagliflozin + Linagliptin low dose (Experimental): 1 tablet once daily
  Interventions: Drug: Empagliflozin + Linagliptin
- Empagliflozin + Linagliptin high dose (Experimental): 1 tablet once daily
  Interventions: Drug: Empagliflozin + Linagliptin

INTERVENTIONS:
Drug: Linagliptin — tablet
  Arms: Linagliptin
Drug: Empagliflozin + Linagliptin — Fixed dose combination.
  Arms: Empagliflozin + Linagliptin low dose
Drug: Empagliflozin + Linagliptin — Fixed dose combination
  Arms: Empagliflozin + Linagliptin low dose
Drug: Empagliflozin + Linagliptin — Fixed dose combination
  Arms: Empagliflozin + Linagliptin high dose
Drug: Empagliflozin placebo + Linagliptin placebo — Matching Empagliflozin + Linagliptin low dose
  Arms: Linagliptin
Drug: Empagliflozin + Linagliptin — Fixed dose combination.
  Arms: Empagliflozin + Linagliptin high dose

SUMMARY:
This trial compare the use of two different doses of Empagliflozin to placebo, in T2DM patients on 16 wks linagliptin treatment and metformin background therapy.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus.
2. Male and female patients on diet and exercise regimen, pre-treated with immediate release metformin for at least 12 weeks, and patients should be on a dose higher or equal to 1500 mg/day of metformin, or maximum tolerated dose, or maximum dose as per local label.
3. HbA1c higher or equal to 8.0% and lower or equal to 10.5% at screening visit.
4. Age 18 years or more at screening.
5. Body Mass Index lower or equal to 45 kg/m2 at screening visit.
6. Signed and dated written informed consent.

Exclusion criteria:

1. Uncontrolled hyperglycemia with glucose level above 270 mg/dl (above 15 mmol/dl) after an overnight fast.
2. Use of any other antidiabetic drug (except metformin background therapy).
3. Acute coronary syndrome, stroke or TIA within 3 months prior to informed consent.
4. Indication of liver disease.
5. Impaired renal function.
6. Gastrointestinal surgery.
7. Treatment with anti-obesity drugs within 3 months prior to screening, or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen, etc.) leading to unstable body weight.
8. Current treatment with systemic steroids at time of informed consent or uncontrolled endocrine disorder except type 2 diabetes mellitus.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 607 (Actual)
Dates: Start 2013-02-08 (Actual); Primary Completion 2015-03-23 (Actual); Study Completion 2015-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (90):
- United States (28):
  - 1275.9.01013 Boehringer Ingelheim Investigational Site, Gulf Shores, Alabama
  - 1275.9.01009 Boehringer Ingelheim Investigational Site, Norwalk, California
  - 1275.9.01015 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1275.9.01017 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1275.9.01011 Boehringer Ingelheim Investigational Site, Northglenn, Colorado
  - 1275.9.01010 Boehringer Ingelheim Investigational Site, Coral Gables, Florida
  - 1275.9.01004 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1275.9.01006 Boehringer Ingelheim Investigational Site, Oldsmar, Florida
  - 1275.9.01001 Boehringer Ingelheim Investigational Site, Palm Coast, Florida
  - 1275.9.01027 Boehringer Ingelheim Investigational Site, Port Orange, Florida
  - 1275.9.01029 Boehringer Ingelheim Investigational Site, Blue Ridge, Georgia
  - 1275.9.01003 Boehringer Ingelheim Investigational Site, Marietta, Georgia
  - 1275.9.01022 Boehringer Ingelheim Investigational Site, Savannah, Georgia
  - 1275.9.01031 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1275.9.01019 Boehringer Ingelheim Investigational Site, Methuen, Massachusetts
  - 1275.9.01024 Boehringer Ingelheim Investigational Site, Troy, Michigan
  - 1275.9.01023 Boehringer Ingelheim Investigational Site, St Louis, Missouri
  - 1275.9.01002 Boehringer Ingelheim Investigational Site, Omaha, Nebraska
  - 1275.9.01007 Boehringer Ingelheim Investigational Site, Newington, New Hampshire
  - 1275.9.01016 Boehringer Ingelheim Investigational Site, Asheboro, North Carolina
  - 1275.9.01025 Boehringer Ingelheim Investigational Site, Burlington, North Carolina
  - 1275.9.01014 Boehringer Ingelheim Investigational Site, Shelby, North Carolina
  - 1275.9.01028 Boehringer Ingelheim Investigational Site, Winston-Salem, North Carolina
  - 1275.9.01018 Boehringer Ingelheim Investigational Site, Dayton, Ohio
  - 1275.9.01005 Boehringer Ingelheim Investigational Site, Corvallis, Oregon
  - 1275.9.01032 Boehringer Ingelheim Investigational Site, Corpus Christi, Texas
  - 1275.9.01030 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1275.9.01021 Boehringer Ingelheim Investigational Site, San Antonio, Texas
- Australia (6):
  - 1275.9.61009 Boehringer Ingelheim Investigational Site, Liverpool, New South Wales
  - 1275.9.61001 Boehringer Ingelheim Investigational Site, St Leonards, New South Wales
  - 1275.9.61003 Boehringer Ingelheim Investigational Site, Carina Heights, Queensland
  - 1275.9.61002 Boehringer Ingelheim Investigational Site, Herston, Queensland
  - 1275.9.61006 Boehringer Ingelheim Investigational Site, Malvern, Victoria
  - 1275.9.61007 Boehringer Ingelheim Investigational Site, Nedlands, Western Australia
- Brazil (5):
  - 1275.9.55002 Boehringer Ingelheim Investigational Site, Brasília
  - 1275.9.55005 Boehringer Ingelheim Investigational Site, Goiânia
  - 1275.9.55001 Boehringer Ingelheim Investigational Site, São Paulo
  - 1275.9.55003 Boehringer Ingelheim Investigational Site, São Paulo
  - 1275.9.55004 Boehringer Ingelheim Investigational Site, São Paulo
- Canada (6):
  - 1275.9.01101 Boehringer Ingelheim Investigational Site, Burnaby, British Columbia
  - 1275.9.01103 Boehringer Ingelheim Investigational Site, Victoria, British Columbia
  - 1275.9.01105 Boehringer Ingelheim Investigational Site, Cornwall, Ontario
  - 1275.9.01106 Boehringer Ingelheim Investigational Site, Hamilton, Ontario
  - 1275.9.01104 Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - 1275.9.01102 Boehringer Ingelheim Investigational Site, Waterloo, Ontario
- 1275.9.34008 Boehringer Ingelheim Investigational Site, Barcelona, El Salvador
- France (7):
  - 1275.9.33006 Boehringer Ingelheim Investigational Site, Bourg-des-Comptes
  - 1275.9.33008 Boehringer Ingelheim Investigational Site, Dessenheim
  - 1275.9.33003 Boehringer Ingelheim Investigational Site, La Riche
  - 1275.9.33012 Boehringer Ingelheim Investigational Site, Paris
  - 1275.9.33002 Boehringer Ingelheim Investigational Site, Saint-Avertin
  - 1275.9.33005 Boehringer Ingelheim Investigational Site, Savonnières
  - 1275.9.33004 Boehringer Ingelheim Investigational Site, Tours
- New Zealand (8):
  - 1275.9.64005 Boehringer Ingelheim Investigational Site, Auckland, New Zealand
  - 1275.9.64006 Boehringer Ingelheim Investigational Site, Auckland, New Zealand
  - 1275.9.64008 Boehringer Ingelheim Investigational Site, Birkenhead Auckland
  - 1275.9.64007 Boehringer Ingelheim Investigational Site, Christchurch Central
  - 1275.9.64004 Boehringer Ingelheim Investigational Site, Christchurch, New Zealand
  - 1275.9.64002 Boehringer Ingelheim Investigational Site, Otahuhu Auckland
  - 1275.9.64001 Boehringer Ingelheim Investigational Site, Takapuna Auckland
  - 1275.9.64003 Boehringer Ingelheim Investigational Site, Tauranga, New Zealand
- Norway (5):
  - 1275.9.47001 Boehringer Ingelheim Investigational Site, Bergen
  - 1275.9.47002 Boehringer Ingelheim Investigational Site, Oslo
  - 1275.9.47003 Boehringer Ingelheim Investigational Site, Oslo
  - 1275.9.47007 Boehringer Ingelheim Investigational Site, Oslo
  - 1275.9.47006 Boehringer Ingelheim Investigational Site, Svelvik
- South Korea (9):
  - 1275.9.82006 Boehringer Ingelheim Investigational Site, Daejeon
  - 1275.9.82009 Boehringer Ingelheim Investigational Site, Deagu
  - 1275.9.82002 Boehringer Ingelheim Investigational Site, Goyang
  - 1275.9.82004 Boehringer Ingelheim Investigational Site, Seongnam
  - 1275.9.82001 Boehringer Ingelheim Investigational Site, Seoul
  - 1275.9.82005 Boehringer Ingelheim Investigational Site, Seoul
  - 1275.9.82007 Boehringer Ingelheim Investigational Site, Seoul
  - 1275.9.82008 Boehringer Ingelheim Investigational Site, Seoul
  - 1275.9.82010 Boehringer Ingelheim Investigational Site, Seoul
- Spain (9):
  - 1275.9.34011 Boehringer Ingelheim Investigational Site, A Coruña
  - 1275.9.34009 Boehringer Ingelheim Investigational Site, Alicante
  - 1275.9.34005 Boehringer Ingelheim Investigational Site, Badía Del Vallès - Barcelona
  - 1275.9.34001 Boehringer Ingelheim Investigational Site, Barcelona
  - 1275.9.34003 Boehringer Ingelheim Investigational Site, Barcelona
  - 1275.9.34004 Boehringer Ingelheim Investigational Site, Barcelona
  - 1275.9.34002 Boehringer Ingelheim Investigational Site, Seville
  - 1275.9.34010 Boehringer Ingelheim Investigational Site, Valencia
  - 1275.9.34006 Boehringer Ingelheim Investigational Site, Vic
- Taiwan (6):
  - 1275.9.88606 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1275.9.88607 Boehringer Ingelheim Investigational Site, Kaohsiung City
  - 1275.9.88602 Boehringer Ingelheim Investigational Site, New Taipei City
  - 1275.9.88603 Boehringer Ingelheim Investigational Site, Taichung
  - 1275.9.88604 Boehringer Ingelheim Investigational Site, Taichung
  - 1275.9.88605 Boehringer Ingelheim Investigational Site, Tainan

REFERENCES:
- [Derived] Softeland E, Meier JJ, Vangen B, Toorawa R, Maldonado-Lutomirsky M, Broedl UC. Empagliflozin as Add-on Therapy in Patients With Type 2 Diabetes Inadequately Controlled With Linagliptin and Metformin: A 24-Week Randomized, Double-Blind, Parallel-Group Trial. Diabetes Care. 2017 Feb;40(2):201-209. doi: 10.2337/dc16-1347. Epub 2016 Dec 2. PMID 27913576
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 16-week open-label (OL) lina 5 period followed by a 1-week OL period with additional placebo administration preceded randomisation to double-blind treatment. Patients were randomised to double blind treatment only when they had not met glycaemic control criteria after the 16-week OL period. All treatments were administered in addition to metformin.
Groups:
- Empagliflozin 25 mg: Patients received 1 fixed dose combination (FDC) Empagliflozin (empa) 25/lina 5 mg tablet and two placebo tablet (1 matching placebo tablet to lina 5 and 1 matching placebo tablet to FDC empa 10/lina 5), administered orally, once every day for 24 weeks during the double blind treatment period.
- Empagliflozin 10 mg: Patients received 1 FDC empa 10/lina 5 mg tablet and two placebo tablet (1 matching placebo tablet to lina 5 and 1 matching placebo tablet to FDC empa 25/lina 5), administered orally, once every day for 24 weeks during the double blind treatment period.
- Placebo: Patients received 1 lina 5 mg tablet and two placebo tablet (1 matching placebo tablet to FDC empa 25/lina 5 and 1 matching placebo tablet to FDC empa 10/lina 5), administered orally, once every day for 24 weeks during the double blind treatment period.
- Linagliptin 5 mg: Patients received 5mg dose of Linagliptin (lina 5), administered orally, once daily for 16 weeks during the OL treatment period, thereafter patients received 1 matching placebo tablet to FDC empa 25/lina 5, and 1 matching placebo tablet to FDC empa 10/lina 5 per day in addition to lina 5 OL, for 1 week during the open-label placebo add-on treatment period.
Period: Open-Label Period
Arm/Group | Empagliflozin 25 mg | Empagliflozin 10 mg | Placebo | Linagliptin 5 mg
Started | 0 | 0 | 0 | 606
Completed | 0 | 0 | 0 | 333
Not Completed | 0 | 0 | 0 | 273
Not completed — Adverse Event | 0 | 0 | 0 | 9
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 13
Not completed — Lost to Follow-up | 0 | 0 | 0 | 14
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 12
Not completed — Other Reasons | 0 | 0 | 0 | 224
Period: Double-Blind Period
Arm/Group | Empagliflozin 25 mg | Empagliflozin 10 mg | Placebo | Linagliptin 5 mg
Started | 111 | 112 | 110 | 0
Completed | 106 | 103 | 105 | 0
Not Completed | 5 | 9 | 5 | 0
Not completed — Adverse Event | 0 | 3 | 2 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 2 | 4 | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — Not treated | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The treated set (TS) consisted of all patients who were randomised and treated with at least 1 dose of study drug during the double-blind part of the trial.
Groups:
- Empagliflozin 25 mg: Patients received 1 FDC Empagliflozin (empa) 25/lina 5 mg tablet and two placebo tablet (1 matching placebo tablet to lina 5 and 1 matching placebo tablet to FDC empa 10/lina 5), administered orally, once every day for 24 weeks during the double blind treatment period.
- Total: Total of all reporting groups
Arm/Group | Empagliflozin 25 mg | Empagliflozin 10 mg | Placebo | Total
Number analyzed (Participants) | 110 | 112 | 110 | 332
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.4 (9.9) | 54.3 (9.5) | 55.9 (9.6) | 55.2 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 46 | 49 | 134
  Male | 71 | 66 | 61 | 198

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline After 24 Weeks Double-blind Randomized Treatment
Description: Change from baseline in Glycated haemoglobin (HbA1c) [%] after 24 weeks of treatment with double-blind trial medication. Baseline was defined as the last observation before the first intake of any double-blind randomised trial medication. The term 'baseline' was not used to refer to measurements before the administration of open-label medication.
Time Frame: Baseline and 24 weeks
Population: The full analysis set (FAS) consisted of all patients in the treated set (TS) who had a baseline HbA1c assessment and at least 1 on-treatment HbA1c assessment during the double-blind part of the trial. Observed Case (OC): In the OC analysis, values after the use of rescue medication were set to missing.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Empagliflozin 25 mg | Empagliflozin 10 mg | Placebo
Number analyzed (Participants) | 110 | 109 | 106
Percentage of HbA1c | -0.56 (0.08) | -0.65 (0.08) | 0.14 (0.09)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg vs Placebo; Superiority of Empagliflozin 25 mg vs. placebo: change in HbA1c using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. Model includes baseline HbA1c as linear covariate(s) & baseline Estimated glomerula filtration rate (eGFR), geographical region, treatment, visit, visit by treatment interaction as fixed effect(s); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -0.70, 95% CI [-0.93 to -0.46], Standard Error of Mean 0.12 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as Empagliflozin 25 mg minus Placebo
Statistical Analysis 2: Comparison: Empagliflozin 10 mg vs Placebo; Superiority of Empagliflozin 10 mg vs. placebo: change in HbA1c using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. Model includes baseline HbA1c as linear covariate(s) & baseline Estimated glomerula filtration rate (eGFR), geographical region, treatment, visit, visit by treatment interaction as fixed effect(s); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -0.79, 95% CI [-1.02 to -0.55], Standard Error of Mean 0.12 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as Empagliflozin 10 mg minus Placebo

2. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline After 24 Weeks of Double-blind Treatment.
Description: Change from baseline FPG (mmol/L) after 24 weeks of treatment with double-blind trial medication.
Time Frame: Baseline and 24 weeks
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | Empagliflozin 25 mg | Empagliflozin 10 mg | Placebo
Number analyzed (Participants) | 109 | 109 | 106
mmol/L | -1.75 (0.18) | -1.46 (0.18) | 0.34 (0.19)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg vs Placebo; Superiority of Empagliflozin 25 mg vs. placebo: change in FPG using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. Model includes baseline FPG, baseline HbA1c as linear covariate(s) & baseline eGFR, geographical region, treatment, visit, visit by treatment interaction as fixed effect(s); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -2.09, 95% CI [-2.61 to -1.57], Standard Error of Mean 0.26 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as Empagliflozin 25 mg minus Placebo
Statistical Analysis 2: Comparison: Empagliflozin 10 mg vs Placebo; Superiority of Empagliflozin 10 mg vs. placebo: change in FPG using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. Model includes baseline FPG, baseline HbA1c as linear covariate(s) & baseline eGFR, geographical region, treatment, visit, visit by treatment interaction as fixed effect(s); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -1.80, 95% CI [-2.31 to -1.28], Standard Error of Mean 0.26 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as Empagliflozin 10 mg minus Placebo

3. Secondary Outcome: Body Weight Change From Baseline After 24 Weeks of Double-blind Treatment
Description: Change from baseline Body weight after 24 weeks of treatment with double-blind trial medication.
Time Frame: Baseline and 24 weeks
Population: FAS (OC)
Measure: Least Squares Mean (Standard Error); unit: kg
Arm/Group | Empagliflozin 25 mg | Empagliflozin 10 mg | Placebo
Number analyzed (Participants) | 110 | 109 | 106
kg | -2.52 (0.25) | -3.06 (0.25) | -0.30 (0.26)
Statistical Analysis 1: Comparison: Empagliflozin 25 mg vs Placebo; Superiority of Empagliflozin 25 mg vs. placebo: change in body weight using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. Model includes baseline weight, baseline HbA1c as linear covariate(s) & baseline eGFR, geographical region, treatment, visit, visit by treatment interaction as fixed effect(s); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -2.22, 95% CI [-2.92 to -1.52], Standard Error of Mean 0.36 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as Empagliflozin 25 mg minus Placebo
Statistical Analysis 2: Comparison: Empagliflozin 10 mg vs Placebo; Superiority of Empagliflozin 10 mg vs. placebo:change in body weight using a restricted maximum likelihood (REML)- based mixed model repeated measures (MMRM) approach. Model includes baseline weight, baseline HbA1c as linear covariate(s) & baseline eGFR, geographical region, treatment, visit, visit by treatment interaction as fixed effect(s); Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; The unstructured covariance structure has been used to fit the mixed model; Mean Difference (Final Values) = -2.77, 95% CI [-3.47 to -2.07], Standard Error of Mean 0.36 — Mean Difference (Final Values) is actually the Adjusted mean difference calculated as Empagliflozin 10 mg minus Placebo

ADVERSE EVENTS:
Time Frame: From first drug administration until 7 days after the last drug administration, up to 126 days (open label treatment period) and 176 days (double blind treatment period).
Arm/Group | Empagliflozin 25 mg | Empagliflozin 10 mg | Placebo | Linagliptin 5 mg
Serious Adverse Events (participants affected / at risk) | 4/110 | 5/112 | 10/110 | 18/606
Other Adverse Events (participants affected / at risk) | 11/110 | 19/112 | 34/110 | 78/606
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 25 mg (N=110) | Empagliflozin 10 mg (N=112) | Placebo (N=110) | Linagliptin 5 mg (N=606)
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
Abscess (Infections and infestations) | 0 | 0 | 0 | 1
Diarrhoea infectious (Infections and infestations) | 0 | 0 | 0 | 1
Erysipelas (Infections and infestations) | 0 | 0 | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1
Pharyngitis bacterial (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 1 | 0 | 0 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cervical radiculopathy (Nervous system disorders) | 0 | 0 | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 0 | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 1
Major depression (Psychiatric disorders) | 0 | 0 | 0 | 1
Mania (Psychiatric disorders) | 0 | 0 | 1 | 0
Calculus ureteric (Renal and urinary disorders) | 1 | 0 | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 1 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 25 mg (N=110) | Empagliflozin 10 mg (N=112) | Placebo (N=110) | Linagliptin 5 mg (N=606)
Nasopharyngitis (Infections and infestations) | 4 | 5 | 8 | 25
Urinary tract infection (Infections and infestations) | 3 | 8 | 7 | 28
Lipase increased (Investigations) | 3 | 4 | 6 | 10
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1 | 7 | 6
Headache (Nervous system disorders) | 2 | 3 | 8 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.